CLINICAL TRIAL: NCT06579586
Title: The Relationship Between Parental Anxiety and Postoperative Pain and Complications in Children Undergoing Tonsillectomy ± Adenoidectomy
Brief Title: Parental Anxiety and Postoperative Pain and Complications in Children Undergoing Tonsillectomy ± Adenoidectomy
Status: Completed | Type: Observational
Sponsor: Sumeyra DOLUOGLU (Other)
Responsible Party: Sponsor-Investigator, Sumeyra DOLUOGLU, Principal Investigator, Saglik Bilimleri Universitesi
Organization: Saglik Bilimleri Universitesi (Other)
Other Study IDs: SumeyraDoluoglu1
Record Dates: First submitted 2024-08-21; First posted 2024-08-30 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Parents; Anxiety; Complication of Surgical Procedure; Pain
Keywords: Parental anxiety; Tonsillectomy; Postoperative pain; Complication of tonsillectomy
MeSH Terms: conditions — Anxiety Disorders; Pain; Pain, Postoperative | interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children undergoing tonsillectomy ± adenoidectomy: It is aimed to understand whether high parental anxiety leads to increased pain in children undergoing tonsillectomy ± adenoidectomy surgery and whether it increases the development of complications.
  Interventions: Behavioral: Survey study

INTERVENTIONS:
Behavioral: Survey study — The Parent's State and Trait Anxiety Inventory (STAI), Anxiety Sensitivity Index-3 (AS-3), and Pain Catastrophising Scale for Parents (PPS-PPS) were completed one day before the operation to measure anxiety level.

SUMMARY:
It is aimed to understand whether high parental anxiety leads to increased pain in children undergoing tonsillectomy ± adenoidectomy surgery and whether it increases the development of complications.

ELIGIBILITY:
Inclusion Criteria:

* 4-15 years old child patient
* Willingness to participate in the study by the patient and/or parent
* No history of psychiatric-mental illness or drug use in the patient and/or parents
* The patient has no craniofacial anomaly, genetic disorder, cleft palate-lip anomaly
* No bleeding disorder or disease

Exclusion Criteria:

* <4 years old, >15 years old paediatric patients
* Not wanting to participate in the study at any stage of the study
* History of psychiatric-mental illness or drug use in the patient and parents
* The patient has craniofacial anomaly, genetic disorder, cleft palate-lip anomaly
* Having a bleeding disorder or disease

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients aged 4-15 years, who had no history of psychiatric-mental illness or drug use in themselves or their parents, and who underwent tonsillectomy + adenoidectomy for chronic tonsillitis or sleep-disordered breathing were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Evaluation the relationship between parents' anxiety level in the preoperative period and pain perception and complications in children undergoing tonsillectomy ± adenoidectomy | 14 days
  Pain perception in parents with high anxiety level and in children of these parents who underwent an operation such as adenotonsillectomy that may cause intense pain sensation was questioned by the parent and then by the child at postoperative 6th hour, 24th hour, 1st week and 2nd week.
Determination of preoperative anxiety level in parents of children undergoing tonsillectomy +/- adenoidectomy with State-Trait Anxiety Inventory | 21 days
  It is a scale consisting of two stages as state and trait anxiety levels. It consists of 40 questions in total, 20 questions each. State anxiety is used to define the level of anxiety in a particular situation, whereas trait anxiety is used to define the anxiety experienced independently of the situation the person is in. Each question is evaluated on a scale of at least 1 (never) and at most 4 points (always) and is expressed in scores ranging from 20-80 points. High scores indicate high levels of anxiety.
Determination of preoperative anxiety level in parents of children undergoing tonsillectomy +/- adenoidectomy with Anxiety Sensitivity Index-3 | 21 days
  Anxiety sensitivity (AS) is characterised as 'an excessive fear of anxiety-related sensations and symptoms that are believed to have harmful physical and/or social consequences'. People with high AS tend to misinterpret sudden, relatively severe and unexplained physical symptoms of anxiety as dangerous, but often tend to avoid them. While '0' means very little, '4' means very much. The score that can be obtained from the scale is between 0-72. The practitioners are asked to indicate to what extent they agree with the statements in each item by taking into account their previous experiences related to the statements in each item, or if they have no experience with that item, they are asked to indicate how they would feel if they experienced that situation. There are no reverse items in the scale. A high score indicates high anxiety sensitivity.
Determination of preoperative anxiety level in parents of children undergoing tonsillectomy +/- adenoidectomy with Pain Catastrophising Scale for Parents | 21 days
  Pain catastrophising is the tendency to over-focus on and exaggerate the response to painful stimuli and their threat value, and to feel more helpless about the pain experience. It was developed because of the need to relate the degree to which parents catastrophise their children's suffering and the effects on their children's well-being and behaviour. It is assessed with a 5-point scale ranging from 0 (not at all) to 4 (very much). Items from the subscales are added to obtain a total score between 0 and 52; higher scores reflect higher levels of catastrophic thinking in parents.

CONTACTS AND LOCATIONS:
Overall Officials: Sumeyra Doluoglu, MD, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Doluoglu S, Gazeloglu AZ, Kocyigit Y, Vural Camalan B, Ozlugedik S. Effects of Parental Anxiety on the Postoperative Pain and Complications of Children Undergoing Adenotonsillectomy. Laryngoscope. 2025 Sep;135(9):3422-3429. doi: 10.1002/lary.32217. Epub 2025 May 5. PMID 40323129